CLINICAL TRIAL: NCT04292522
Title: Care Pathway for Children With Autism Spectrum Disorder Included in the ELENA Cohort : Matching to the National Health Data System
Brief Title: Care Pathway for Children With Autism Spectrum Disorder Included in the ELENA Cohort
Acronym: ELENA-SNDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0443-UF7969
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Care pathway; Health administrative database
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autism Spectrum Disorder (ASD) is lifelong neurodevelopmental disorder that affect social communication and interaction and includes limited and repetitive patterns of behavior (DSM 5). In France, national guidelines about practices recommends early and specific interventions but care pathway are not well described for ASD children. The national health insurance information system record demographic data, medical condition, and reimbursed drug over 98% of the French population. In addition, the ELENA cohort is a large cohort of children with ASD followed for 6 years. Data collected include clinical characteristics of children (IQ, severity of ASD...) and parents (educational level, professional status...).

The first objective of this project is to identify patterns of care trajectories using data from ELENA cohort matched to data from national health insurance information system. Secondary objectives are to examine the links between patterns of care trajectories and clinical characteristics, social environment of autistic children.

ELIGIBILITY:
Inclusion criteria:

- Included in ELENA Cohort

Exclusion criteria:

- Opposable to reuse data

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with ASD included in the ELENA Cohort
Sampling Method: Probability Sample
Enrollment: 903 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Care pathway | 1 day
  Care pathway will be built from administrative database from birth to 2019
Clinical characteristics | 1 day
  Clinical, social and environmental data of children from ELENA cohort

CONTACTS AND LOCATIONS:
Overall Officials: Amaria Baghdadli, Professor, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC